CLINICAL TRIAL: NCT02375009
Title: Glaucoma Management in the African-Derived Developing World Using Trabeculoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Anthony Realini, Associate Professor of Ophthalmology, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1411505682
Record Dates: First submitted 2015-01-26; First posted 2015-03-02 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Cohort (Experimental): All subjects will receive bilateral 360 degree Selective Laser Trabeculoplasty therapy in a single session, but will be randomized to one of three treatment sessions at times 0, Month 3 and Month 6. Subjects will be washed out of current IOP-lowering therapy 4-6 weeks pre-SLT. Subjects continuing on meds beyond time 0 will provide a comparator to early SLT to quantify regression to the mean.
  Interventions: Procedure: Selective laser trabeculoplasty

INTERVENTIONS:
Procedure: Selective laser trabeculoplasty — laser therapy to trabecular outflow pathway of the eye to lower intraocular pressure, delivered to 360 degrees of both eyes in a single session

SUMMARY:
This proposal aims to evaluate selective laser trabeculoplasty (SLT) as a safe and effective therapy to control open-angle glaucoma and reduce the risk of progression to visual dysfunction or blindness in the African-derived developing world. If funded, this work will complete the characterization of SLT's safety and efficacy profile as a means of long-term disease control in this population. This work will support the translation of SLT into a structured public health initiative to reduce glaucoma-related vision loss throughout the African-derived developing world.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of blindness in the African-derived developing world and represents a significant public health challenge as the disease burden is substantial. In Ghana, the prevalence of open-angle glaucoma over age 40 is 8.5%. In Barbados, the prevalence is 7.0%. In neighboring St. Lucia, the prevalence has been estimated at 8.8% with a 16% ten-year incidence of glaucoma-related blindness in one or both eyes. (In contrast, the prevalence in US adults is 1.9%.) The burden of glaucoma-related visual dysfunction is also substantial in the developing world. Because the application of medical and surgical therapies is limited by issues such as cost, availability, and limited regional surgical expertise, undertreatment is pervasive. Also, there is little access to low vision or vision rehabilitation services and minimal social support for the visually impaired. Laser trabeculoplasty may be a part of the solution to the developing world's burgeoning glaucoma burden. The treatment is fast, safe, minimally invasive and requires minimal post-treatment care; the equipment is portable; and the incremental cost of trabeculoplasty treatment is small once the equipment and expertise are on-site. Our recent study in St. Lucia demonstrated that laser trabeculoplasty lowers IOP by an amount likely to favorably alter the clinical course of glaucoma (versus no treatment) and has the potential to bend the glaucoma-related blindness curve in the African-derived developing world. Our long-term goal is to translate this finding through a public health initiative by establishing a pan-Caribbean glaucoma laser program to provide safe, effective, and cost-effective therapy for glaucoma in this underserved and overburdened region. Before this can happen, several important research questions remain unanswered regarding SLT in this population and comprise the specific aims of this proposal. What is the long-term efficacy of SLT in this population? Is repeat SLT effective once the IOP reduction of initial SLT wanes? Are the results obtained in St. Lucia generalizable to other developing nations populated by people of African descent? In this application, we propose a prospective cohort study in St. Lucia in which qualifying subjects with open-angle glaucoma will receive bilateral selective laser trabeculoplasty, will be followed to failure of initial SLT, and will undergo repeat SLT and again be followed to failure. The long-term safety and efficacy of both initial and repeat SLT in glaucoma patients of African descent will thus be established. Further, we will replicate the cohort study in Dominica to confirm external validity of the St. Lucia outcomes. This proposal is designed to answer the questions posed above and thus to complete the research phase of this project and facilitate translation of the research findings into the public health space. Considering the population of the African-derived developing world, the prevalence of glaucoma in this population, and the observed preliminary benefits of laser therapy, this project's output could ultimately reduce the risk of glaucoma-related visual dysfunction in hundreds of thousands of individuals throughout the developing world.

ELIGIBILITY:
Inclusion Criteria:

* Afro-Caribbean ancestry
* Ages 30 and above
* Open-angle glaucoma (ISGEO criteria)
* CDR≥0.7 or CDR asymmetry ≥0.2 or rim width ≤0.1 CDR with typical VF loss; or
* CDR≥0.8 or CDR asymmetry ≥0.3 (if unable to get VF); or
* VA <20/400 and IOP ≥ 32 mmHg (if unable to get VF or CDR)
* Receiving ≤2 topical IOP-lowering medications
* IOP between 17-35 mmHg in both eyes after 30-day washout

Exclusion Criteria:

* Any glaucoma other than open-angle glaucoma
* Advanced glaucoma (CDR > 0.9 or field loss in central 10º)
* History of:
* Prior glaucoma laser or surgery
* Ocular inflammation within 3 months
* Ocular trauma or intraocular surgery within 6 months

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Probability of 12-month success (Proportion of subjects with 20% or greater IOP reduction 12 months following SLT) | 12 months
  Proportion of subjects with 20% or greater IOP reduction 12 months following SLT
Repeat probability of 12-month success (Proportion of subjects with 20% or greater IOP reduction from baseline 12 months after repeat SLT) | 12 months after as-needed repeat SLT
Generalizability of IOP-lowering efficacy to populations other than St. Lucia (significance of a site term in a predictive model of IOP reduction) | 12 months
  Evaluate significance of a site term in a predictive model of IOP reduction following SLT to determine if response to IOP is site dependent

SECONDARY OUTCOMES:
Median survival time following initial SLT (Time from initial SLT to when 50% of subjects no longer manifest a 20% or greater reduction in IOP from baseline) | Through up to five years of follow-up
  Time from initial SLT to when 50% of subjects no longer manifest a 20% or greater reduction in IOP from baseline
Mean IOP reduction (Descriptive analysis of mean (+/- SD) IOP reductions from baseline) | through up to five years of follow-up
  Descriptive analysis of mean (+/- SD) IOP reductions from baseline at each 12-month period following initial and repeat SLT, separately

CONTACTS AND LOCATIONS:
Overall Officials: Tony Realini, MD, MPH, Principal Investigator — West Virginia University Eye Institute
Locations (1):
- West Virginia University Eye Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Realini T, Shillingford-Ricketts H, Burt D, Balasubramani GK. Clinical outcomes following selective laser trabeculoplasty in Afro-Caribbean patients with glaucoma at high risk for progression. Br J Ophthalmol. 2022 Sep;106(9):1235-1239. doi: 10.1136/bjophthalmol-2020-317117. Epub 2021 Apr 9. PMID 33836987
- [Derived] Realini T, Shillingford-Ricketts H, Burt D, Balasubramani GK. West Indies Glaucoma Laser Study (WIGLS)-2: Predictors of Selective Laser Trabeculoplasty Efficacy in Afro-Caribbeans With Glaucoma. J Glaucoma. 2018 Oct;27(10):845-848. doi: 10.1097/IJG.0000000000001018. PMID 29965865